#### **COVER PAGE**

#### STATISTICAL ANALYSIS PLAN

November 2, 2017

Final Version 1.0

NCT03178942

A Randomized, Double-Blind, Parallel-Design, Multiple-Site Study to Evaluate the Therapeutic Equivalence of Permethrin Cream, 5% (Encube Ethicals) Compared to Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.) in the Treatment of Scabies

Protocol Number: 71675502 Novum Study Number: 71675502

Permethrin Cream, 5%

Protocol / Study No. 71675502

#### STATISTICAL ANALYSIS PLAN

A Randomized, Double-Blind, Parallel-Design, Multiple-Site Study to Evaluate the Therapeutic Equivalence of Permethrin Cream, 5% (Encube Ethicals) Compared to Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.) in the Treatment of Scabies

Protocol Number: 71675502 Novum Study Number: 71675502

#### **Sponsor:**

Encube Ethicals Unit No. 24, Steelmade Indl Estate, Opposite To Jalaram Store, Marol, Andheri East, Mumbai, Maharashtra 400059, India

#### **Contract Research Organization:**

Novum Pharmaceutical Research Services 225 W. Station Square Drive, Suite 200 Pittsburgh, PA 15219

November 2, 2017

Final Version 1.0

#### MONTHM PIDERMACIEL DE AL PEREARCH SERVICES. STATESTICAL ANALYSIS PEAN

Permethrin Crosm, 5%

Protocol / Study No. 7167:5502

#### LAF Final Version Approvals

A Randomized, Double-Blind, Parallel-Design, Multiple-Site Study to Evaluate the Therapeutic Equivalence of Permethrin Cream, 5% (Uncube Ethicals) Compared to Elimite<sup>17st</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.) in the Treatment of Scabies

| Written By: Signature: Jianhua Liu, MSc Senior Biostatistician Novum Pharmaceutical Research Services | Date: 11/14/2017 |
|---|---|
| Reviewed By: Signature: Pina D'Angelo, MS Executive Director, Scientific Affaits (Biostatistics) Novum Pharmaceutical Research Services | Date: NOV 14, 2017 |
| Approved By: Signature: Pratik Kaman GM- Strategy & Commercial | Date: 10/1401/2013- |

Encube Ethicals Pvt Ltd

Permethrin Cream, 5%

Protocol / Study No. 71675502

## **Revision History**

| VERSION | DATE | DESCRIPTION OF REVISIONS | REVISED<br>BY |
|---|---|---|---|
| Draft 1.0 | July 26, 2017 | New Document | Jianhua Liu |
| Final 1.0 | November 2, 2017 | Incorporate client comments and finalize SAP | Jianhua Liu |

#### Permethrin Cream, 5%

Protocol / Study No. 71675502

#### **List of Abbreviations and Definition of Terms**

ADaM Analysis Data Model

AE Adverse Event BP Blood Pressure

C Celsius

CRF Case Report Form

CDISC Clinical Data Interchange Standards Consortium

CRO Contract Research Organization

F Fahrenheit

FDA Food and Drug Administration

HR Heart Rate Hg Mercury

HIV Human Immunodeficiency Virus

ICF Informed Consent Form

ICH International Conference on Harmonization

IND Investigational New Drug

IWRS Interactive Web Response System LOCF Last Observation Carried Forward

MedDRA Medical Dictionary for Regulatory Activities

mITT Modified Intent-to-Treat

LOCF Last Observation Carried Forward OGD The Office of Generic Drugs

PP Per-Protocol

SAE Serious Adverse Event
SAP Statistical Analysis Plan
SAS Statistical Analysis System
SDTM Study Data Tabulation Model
USA United States of America

| Perm | eth | rin | Cream. | 5% |
|---------|------|-------|-----------|---------|
| 1 (1111 | cui. | 1 111 | Ci Caiii. | ., / () |

## Protocol / Study No. 71675502

#### TABLE OF CONTENTS

| 1. | INTRODUCTION | 8 |
|---|---|---|
| | OBJECTIVES | |
| 3. | OVERALL STUDY DESIGN | 8 |
| 4. | RANDOMIZATION AND BLINDING | 11 |
| 5. | SAMPLE SIZE | 11 |
| 6. | STUDY ENDPOINT | 11 |
| 7. | STUDY POPULATIONS | 12 |
| 8. | STATISTICAL ANALYSIS METHODS | 12 |
| | 8.1 Baseline Characteristics | 13 |
| | 8.1.1 Patient Disposition | 13 |
| | 8.1.2 Demographic and Other Baseline Characteristics | 13 |
| | 8.1.3 Medical History | |
| | 8.1.4 Concomitant Medications | 14 |
| | 8.1.5 Pregnancy Test | 14 |
| | 8.2 Efficacy Analyses. | |
| | 8.2.1 Primary Efficacy Analysis | 14 |
| | 8.2.2 Supportive Analyses | |
| | 8.2.3 Treatment-by-Site Interaction and Pooling of Clinical Sites | |
| | 8.3 Safety Analysis | |
| | 8.3.1 Adverse Events | 16 |
| | 8.3.2 Vital Signs | 17 |
| | 8.4 Multiple Comparisons | 17 |
| | 8.5 Methods for Handling Missing Data | 17 |
| | 8.6 Interim Analyses | |
| 9. | TABLE, LISTING AND FIGURE SHELLS | 17 |
| | T14.1.1 Summary of Patient's Disposition | |
| | T14.1.2 Summary of Protocol Deviations | |
| | T14.1.3.1 Summary of Patients Excluded from Efficacy Analysis (Population | |
| | Determination) | 21 |
| | T14.1.3.2 Summary of Patients Included in Analysis Population by Study Center | 22 |
| | T14.1.4 Summary of Demographic Data and Baseline Characteristics (Safety | |
| | Population) | 24 |
| | T14.1.5 Summary of Demographic Data (Per-Protocol Population) | |
| | T14.1.6 Summary of Microscopic Evaluation of Scabies (Per-Protocol Population) | |
| | T14.1.7 Summary of Frequency of Scabies Signs and Symptoms Rating (Per-Protocol | |
| | Population) | 27 |
| | T14.1.8.1 Summary of Equivalence Analysis Results of Primary Efficacy Endpoint | |
| | (Proportion of Patients in each Treatment Group with Therapeutic Cure | |
| | (Parasitological Cure plus Clinical Cure) of Scabies at Day 28 ± 4) (Per-Protocol | |
| | Population) | 28 |
| | 1 / | _ |

## Permethrin Cream, 5%

Protocol / Study No. 71675502

| T14.1.8.2 Sensitivity Analysis Summary of Equivalence Analysis Efficacy Endpoint (Proportion of Patients in each Treatment Therapeutic Cure (Parasitological Cure plus Clinical Cure) of | Group with<br>f Scabies at Day 28 |
|---|---|
| ± 4) (Safety Population)<br>T14.1.9.1 Supportive Analysis #1: Summary of Equivalence Analysis | |
| Primary Efficacy Endpoint (Per-Protocol Population) | |
| T14.1.9.2 Supportive Analysis #2: Summary of Equivalence Analysis | |
| Primary Efficacy Endpoint (Per-Protocol Population) | |
| T14.1.9.3 Supportive Analysis #3: Summary of Equivalence Analysis | |
| Primary Efficacy Endpoint (Per-Protocol Population) | |
| T14.1.10 Summary of Frequency of Patient Pruritus Assessment ( | |
| Population) | • |
| T14.1.11 Overall Summary of Adverse Events | |
| T14.1.12 Summary of Frequency of Adverse Events by Body Syst | |
| Population) | |
| T14.1.13 Summary of Frequency of Adverse Events by Relationsh | |
| Population) | |
| T14.1.14 Summary of Frequency of Adverse Events by Severity ( | |
| T14.1.15 Summary of Frequency of Serious Adverse Events (Safe | |
| T14.1.16 Summary of Vital Signs (Safety Population) | |
| T14.1.17 Summary of Frequency of Patients with Re-Infestation fi | |
| (treatment success) to Day 28 (treatment failure) (Per-Protoco | |
| T14.1.18 Summary of Frequency of Patients who are Therapeutic | |
| ± 4 (Per-Protocol Population) | |
| L16.2.1 Listing of Discontinued Patients | 39 |
| L16.2.2 Listing of Protocol Deviations | |
| L16.2.3 Patients Excluded from the Per-Protocol Population | 41 |
| L16.2.4.1 Listing of Demographic Data | 42 |
| L16.2.4.2 Listing of Medical History | 43 |
| L16.2.4.3 Listing of Concomitant Medication | 44 |
| L16.2.4.4 Listing of Treatment for Family Members/Close Contac | |
| L16.2.5.1 Listing of Visit Date Information | |
| L16.2.5.2 Listing of Drug Administration | 47 |
| L16.2.6.1 Listing of Scabies Signs and Symptoms Rating and Mic | |
| of Scabies | |
| L16.2.6.2 Listing of Patient Pruritus Assessment | |
| L16.2.6.3 Listing of Investigator Evaluator Initials On Scabies Sig | |
| Rating | |
| L16.2.7 Listing of Adverse Events by Treatment | |
| L16.2.8.1 Listing of Pregnancy Test Results | |
| L16.2.8.2 Listing of Vital Signs | |
| F15.1.1 Histogram of Proportion of Patients with Therapeutic Cur | - |
| Reference: | 55 |

Permethrin Cream, 5% Protocol / Study No. 71675502

■ Encube Ethicals■  11/2/2017

#### Permethrin Cream, 5%

Protocol / Study No. 71675502


#### 1. INTRODUCTION

This Statistical Analysis Plan (SAP) is based on the final Clinical Study Protocol 71675502 [Rev 1] dated 10/31/2017. The SAP provides details on the planned statistical methodology for the analysis of the study data. The SAP also outlines the statistical programming specifications for the tables, listings and figures.

This SAP describes the study endpoints, derived variables, anticipated data transformations and manipulations, and other details of the analyses not provided in the study protocol. This SAP therefore outlines in detail all other aspects pertaining to the planned analyses and presentations for this study.

The following documents were reviewed in preparation of this SAP:

- Final Clinical Study Protocol 71675502 [Rev 1] dated 10/31/2017.
- Case Report Form Booklet Version 1.0 for Novum Study No. 71675502

The reader of this SAP is encouraged to also read the clinical protocol for details on the conduct of this study, and the operational aspects of clinical assessments and timing for completing a patient in this study.

#### 2. OBJECTIVES

The objectives of this study are to:

- 1. Evaluate the therapeutic equivalence of the Test formulation, Permethrin Cream, 5% (Encube Ethicals) to the marketed product, Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.) in patients with scabies.
- 2. Compare the safety of Test and Reference treatments in patients with scabies.

#### 3. OVERALL STUDY DESIGN

This randomized, double-blind, parallel-design, multiple-site study is designed to evaluate the therapeutic efficacy and safety of a generic Permethrin Cream, 5% (Encube Ethicals) compared to the FDA Reference Listed Drug (RLD), Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.) in patients with scabies.

Before any study-specific procedures are performed, all patients will read and sign the IRB-approved informed consent that meets all criteria of current FDA and International Conference of Harmonisation (ICH) regulations. For patients who are considered minors in the state the study is being conducted (< 18 years in most states) the parent or legal guardian should sign the consent form and the child will be required to sign a patient "assent" form, as appropriate. Patients 11-17 years of age will read and sign an IRB-approved assent form and patients 6-10

#### Permethrin Cream, 5%

Protocol / Study No. 71675502

years of age will provide verbal assent. Patients 2-5 years of age will be exempt from providing assent based on the child's comprehension and cognitive skills.

Approximately 250 eligible patients, 2 years of age and older with a clinical diagnosis of active scabies based on signs and symptoms and confirmation of microscopic evidence of scabies mites in the skin will be randomized in a 1:1 ratio (Test: Reference) to one of the two study products as follows:

- Test: Permethrin Cream, 5%, (Encube Ethicals)
- Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

Patients will be instructed to self-administer a single dose of study product or, if patient is a child, then parent/guardian will apply study product to him/her on Day 1 according to the dosing instructions provided. A second application may be required if presence of scabies infestation is microscopically demonstrated (i.e., living mites, viable mite eggs, or mite fecal matter present) at Visit 2. The second dose will be self-administered by the patient or if patient is a child, then parent/guardian will apply study product to him/her at Visit 2. Eligible household members and close contacts of the patient will be offered permethrin cream (if they are in need of treatment) as a method to reduce cross-contamination within a household. Additionally, household members will be requested to follow the standard hygiene practices. Patients whose household members are not willing to comply with the standard of care for Scabies management (i.e., use of generic permethrin cream and standard hygiene practices) will not be enrolled in the study.

During the study, patients will visit the clinical center for a total of three scheduled visits:

- Visit 1 (Day 1): Screening/Baseline
- Visit 2 (Day  $14 \pm 4$ ): Interim Visit
- Visit 3 (Day  $28 \pm 4$ ): End of Study or Early Termination

Final assessments will be carried out at Visit 3 (Day  $28 \pm 4$ ), which is the test-of-cure visit. The test-of-cure visit will occur 4 weeks ( $\pm$  4 days) after the end of the single application treatment on study Day 1 or 2 weeks ( $\pm$  4 days) after the end of a second application, if necessary, on study Visit 2. Therapeutic cure of scabies will be evaluated based on microscopic evidence of absence of scabies infestation (i.e., no living mites, no viable mite eggs, and no mite fecal matter), visual evidence of absence of new lesions and healing of original lesions, regardless of the presence of post-scabetic nodules (i.e., post-scabetic nodules need not be considered as new lesions or persistence of old lesions). The primary statistical analysis of interest is the proportion of patients in each treatment group with therapeutic cure (parasitological cure plus clinical cure) of scabies.

## Permethrin Cream, 5%

Protocol / Study No. 71675502

## **Figure 1 Study Schematic**

| | Visit 1 | Visit 2 | Visit 3 |
|---|---|---|---|
| | Screening/Baseline | Interim Visit | (Day $28 \pm 4$ ) |
| | (Day 1) | (Day $14 \pm 4$ ) | End of Study |
| | | | or Early Termination |
| Informed Consent | X | | |
| Medical history and<br>Baseline Demographics | X | | |
| Vital Signs | X | | X |
| Adverse Events | X | X | X |
| Concomitant Medications | X | X | X |
| Microscopic Examination | X | X | X |
| Scabies Signs and Symptoms Rating (pruritus, lesion count) | X | X | X |
| Urine Pregnancy Test | X | | X |
| Review Inclusion/Exclusion Criteria | X | | |
| Collect and Review Diary | | X | X |
| Provide Diary | X | X | |
| Dispense Study Product | X | X* | |
| Collect and Weigh Study<br>Product | | X | X* |

<sup>\*</sup>If retreatment is necessary, the originally dispensed (i.e., at Visit 1) study product will be dispensed at Visit 2 and collected at Visit 3.

#### Permethrin Cream, 5%

Protocol / Study No. 71675502

#### 4. RANDOMIZATION AND BLINDING

The study product will be randomized, packaged and blinded by an independent packaging company. Randomization will be pre-planned according to a computer-generated randomization schedule. All randomized study products will be blinded and packaged in sealed boxes. Each block will contain two patients' worth of product (1 Test and 1 Reference). Each patient kit will include 1 x 60 gram tube of study product, which should be sufficient for full treatment.

The randomization number will be a unique four-digit number. Patient numbers will be assigned immediately before dispensing of study product and in ascending sequential order, beginning with the lowest available number at the study site. Each patient kit and each dispensed study tube should include the four-digit patient number on the label.

At the end of the study, after all the clinical data have been entered and the study database has been locked, a copy of the randomization schedule will be sent to the statistician.

The Investigator, staff at the study site, study monitors, and data analysis/management personnel will be blinded to the patient assignment.

#### 5. SAMPLE SIZE

For the primary endpoint analysis (proportion of patients in the PP population who are considered to be a Therapeutic Cure on Day  $28 \pm 4$ ), sample size is estimated for therapeutic equivalence of the Test to the Reference product.

Based on data from a previous bioequivalence study conducted to support approval of the first generic product of permethrin cream, 5%, the therapeutic cure rate ( $p_R$ ) of the Reference product (Elimite<sup>TM</sup> permethrin cream 5%) is expected to be about 88% in the PP population. Assuming that the Therapeutic Cure rate for the Test group ( $p_T$ ) is an absolute difference of 5% lower than the Reference group (i.e.,  $p_T$ - $p_R$  = -5%), a sample size of 107 patients in each active group in PP population will provide at least 90% power to demonstrate therapeutic equivalence (i.e., the 90% confidence interval [Yates' continuity corrected] on  $p_T$ - $p_R$  is within a defined equivalence range [-20%, +20%]).

To allow for approximately 14 % of patients who may drop out from the study or are otherwise non-evaluable, approximately 250 patients (125 in each treatment group) will be randomized, such that there will be an estimated 214 patients (107 per group) in the PP population for statistical evaluation of therapeutic equivalence.

#### 6. STUDY ENDPOINT

The primary efficacy endpoint is the proportion of patients in each treatment group with Therapeutic Cure (parasitological cure plus clinical cure) of scabies at the test-of-cure visit

#### Permethrin Cream, 5%

Protocol / Study No. 71675502

conducted at Day  $28 \pm 4$ . A parasitological cure is defined as failure to demonstrate microscopically the presence of scabies infestation (i.e., no living mites, no viable mite eggs, and no mite fecal matter present). A clinical cure is defined as visual evidence of absence of new lesions and healing of original lesions, regardless the presence of post-scabietic nodules (i.e., post-scabietic nodules need not be considered as new lesions or persistence of old lesions).

Patients who do not respond to the initial treatment and have new lesions or microscopic confirmation of mites, ova, or fecal matter on Day  $14 \pm 4$  will be treated as treatment failure in the final analysis on Day 28.

#### 7. STUDY POPULATIONS

#### Per-Protocol (PP) Population

The PP population will include:

- Met the inclusion/exclusion criteria as defined in this protocol at Visit 1.
- Did not take any prohibited medications throughout the study.
- Did not have any significant deviations from the protocol. Did not develop any
  concurrent dermatological condition or illness exhibiting symptoms similar to
  scabies, or symptoms that in the Investigator's opinion would interfere with
  endpoint assessments.
- Completed the last study visit (Visit 3) Day  $28 \pm 4$ .

Patients will be included in the PP population as treatment failures in the final analysis on Day 28 (provided they had no significant protocol deviations) if they 1) withdrew from the study because of lack of efficacy, 2) show therapeutic cure at Day  $14 \pm 4$  but re-infestation at Day  $28 \pm 4$ , or 3) do not respond to the initial treatment and have new lesions or microscopic confirmation of mites, ova, or fecal matter on Day  $14 \pm 4$ .

#### **Safety Population**

The safety population will include all patients who are randomized who applied at least one dose of the assigned study product.

#### 8. STATISTICAL ANALYSIS METHODS

If not otherwise specified, statistical significance is defined as p < 0.05 and is two-tailed. Data will be summarized with respect to demographic and baseline characteristics and safety variables.

#### Permethrin Cream, 5%

Protocol / Study No. 71675502

For categorical variables, the number and percentage of each category within a parameter will be calculated for non-missing data. For continuous variables, statistics will include n, mean, standard deviation, median, minimum and maximum values.

All statistical analyses will be conducted using SAS<sup>®</sup>, Version 9.4 or higher. Datasets will be prepared using headings from Clinical Data Interchange Consortium (CDISC), Study Data Tabulation Model (SDTM) implementation for human clinical trials, and ADaM (Analysis Dataset Model).

#### **8.1 Baseline Characteristics**

#### **8.1.1 Patient Disposition**

The patient disposition information will be summarized by treatment. The number of patients randomized, treated with study medication will be tabulated by treatment. In addition, completion status and primary reason for withdrawal will be summarized by treatment.

#### 8.1.2 Demographic and Other Baseline Characteristics

Baseline comparability of all treatment groups will be evaluated separately in the PP and Safety populations.

The following baseline demographics (determined from their initial study visit) will be evaluated:

- Age (years)
- Sex (male/female)
- Ethnicity (Hispanic/non Hispanic)
- Race (White, Black/African American, Native Hawaiian or Other Pacific Islander, Asian, American Indian or Alaska Native, Other)
- Baseline severity score of nocturnal itching
- Severity of lesion count infestation pretreatment (mild, moderate, severe)

Summary tables by treatment will be presented. Continuous variables will be summarized using descriptive statistics (n, mean, standard deviation, median, minimum, maximum). Categorical variables will be summarized using frequencies and percentage.

Baseline comparability of the treatments will be presented using Chi-square test for the categorical variables, and Analysis of Variance for the continuous variables.

All data will be listed by treatment and patient.

#### Permethrin Cream, 5%

Protocol / Study No. 71675502

#### 8.1.3 Medical History

At Visit 1 patients will be questioned about medical history, including acute and chronic medical history and medical history relevant to their scabies.

Medical history data will be listed by treatment and patient.

#### **8.1.4** Concomitant Medications

All concomitant medication use within 6 months of Visit 1 and throughout the study will be recorded.

All prior and concomitant medications taken since screening until the end of the study will be listed by treatment and patient.

## 8.1.5 Pregnancy Test

All females of childbearing potential will have a urine pregnancy test performed at Visit 1 and Visit 3.

Pregnancy test results will be listed by treatment and patient.

#### **8.2 Efficacy Analyses**

#### **8.2.1 Primary Efficacy Analysis**

#### **Bioequivalence with Clinical Endpoints Analysis**

The proportion of patients in each treatment group with Therapeutic Cure is the primary efficacy endpoint of the study.

The Per Protocol (PP) Population will be used for the analysis of equivalence.

Based on the usual method used in OGD for binary outcomes, the 90% confidence interval for the difference in success proportions between test and reference treatment should be contained within [-0.20, +0.20] (or [-20%, +20%] in percent) in order to establish equivalence.

The compound hypothesis to be tested is:

$$H_0: P_T - P_R < -20\% \text{ or } P_T - P_R > 20\% \text{ versus}$$

$$H_A: -20\% \le P_T - P_R \le 20\%$$

#### Permethrin Cream, 5%

Protocol / Study No. 71675502

where  $P_T$  = percent cure rate of test treatment

 $P_R$  = percent cure rate of reference treatment.

Let

 $n_T$  = sample size of test treatment group

 $cn_T$ = number of cured patients in test treatment group

 $n_R$  = sample size of reference treatment group

 $cn_R$ = number of cured patients in reference treatment group

$$\hat{P}_T = c n_T / n_T$$
  $\hat{P}_R = c n_R / n_R$ , and

$$se = (\hat{P}_T (1 - \hat{P}_T)/n_T + (\hat{P}_R (1 - \hat{P}_R)/n_R)^{1/2})$$

where  $\hat{P}_T$  = estimated cure rate (%) of test treatment

 $\hat{P}_R$  = estimated cure rate (%) of reference treatment.

The 90% confidence interval for the absolute difference between the proportions of patients in test and reference who are considered a therapeutic cure (primary) will be calculated as follows:

$$L = (\hat{P}_T - \hat{P}_R) - 1.645 se$$

$$U = (\hat{P}_T - \hat{P}_R) + 1.645 se$$

If the 90% confidence interval<sup>0</sup> for the absolute difference between the proportion of patients who are considered a therapeutic cure (primary) in the Test and Reference groups is contained within the range [-20% + 20%] then bioequivalence of the Test product to the Reference product will be considered to have been demonstrated for the primary endpoint.

#### Sensitivity Analysis for Primary Efficacy Endpoint

As a sensitivity analysis, the primary efficacy analysis will be performed on the safety population using LOCF. This analysis will use LOCF such that subjects with no post-dose data will be considered as non-responders.

#### 8.2.2 Supportive Analyses

The following supportive analyses will be performed for the primary endpoint:

1. The primary analysis will be performed including patients who completed Visit 2 within  $14 \pm 2$  days and Visit 3 within  $28 \pm 4$  days.

#### Permethrin Cream, 5%

Protocol / Study No. 71675502

- 2. The primary analysis will be performed including patients who completed Visit 2 within  $14 \pm 2$  days and Visit 3 between Day 26 and Day 32, inclusive.
- 3. The primary analysis will be performed including patients who completed Visit 2 within  $14 \pm 2$  days and Visit 3 within  $28 \pm 2$  days.

To declare therapeutic equivalence of the Test product to the Reference product, therapeutic equivalence must be demonstrated for only the primary analysis.

#### 8.2.3 Treatment-by-Site Interaction and Pooling of Clinical Sites

As this is a multiple-site study, the interaction of treatment-by-site may be evaluated for the primary efficacy endpoint in the PP population (for equivalence testing). The treatment-by-site interaction will be evaluated by the Breslow-Day test for homogeneity of the odds ratio at the 5% significance level (p < 0.05). A site(s) with a low enrollment rate(s) may be pooled with its geographically closest site, so as to avoid bias in the estimation of a treatment-by-site interaction effect. The pooling will be done for low enrolling sites that account for less than 4-7% of the total number of patients in the PP population at the site with the highest enrolling rate in the PP population. If the treatment-by-site interaction term is found to be statistically significant (p < 0.05) for the primary endpoint, then the interaction term will also be assessed for clinical relevance before pooling the data across sites. This will include examination of Therapeutic Cure rates at each site where sample sizes per treatment may be influential in the assessment of the interaction.

#### 8.3 Safety Analysis

Safety analysis will be conducted on safety population.

#### **8.3.1** Adverse Events

All the adverse events (AEs) reported throughout the study will be coded and classified according to the MedDRA (Medical Dictionary for Regulatory Activities) coding dictionary (Version 20.0 or higher). Each adverse event is to be evaluated for date of start and end, seriousness, severity, causal relationship with the study drugs, action taken and outcome.

All AEs will be listed by treatment and patient.

A summary table of the number and percent of patients with AEs by system organ class, preferred term, and treatment will be presented. Each patient will be counted only once within each preferred term.

#### Permethrin Cream, 5%

Protocol / Study No. 71675502

A frequency summary table of the number of AEs by system organ class, preferred term, severity, and treatment will be presented. Severity will be classified as "Mild", "Moderate", or "Severe".

Similarly, a frequency summary table of the number of AEs by system organ class, preferred term, and relationship to a study drug, and treatment will be presented. Relationship to a study drug will be classified as "Not Related" or "Related".

Adverse event frequencies will be compared between treatments using Fisher's exact test.

#### 8.3.2 Vital Signs

The patient's vital signs will be recorded (heart rate, blood pressure, temperature and respiration rate) at Visit 1 and Visit 3.

Descriptive summaries (number of observations, mean, standard deviation, minimum, median and maximum) will be provided by treatment and visit.

All data will be listed by treatment and patient.

#### **8.4 Multiple Comparisons**

No multiple comparison adjustment will be made in this study.

#### 8.5 Methods for Handling Missing Data

For demographic and baseline characteristics, each variable will be analyzed using all available data. Patients with missing data will be excluded only from analyses for which data are not available.

#### 8.6 Interim Analyses

There is no interim analysis planned in this study.

#### 9. TABLE, LISTING AND FIGURE SHELLS

The following shells are provided in order to provide a framework for the display of data from this study. These shells may not be reflective of every aspect of this study but are intended to show the general layout of the Tables, Listings and Figures that will be included in the final clinical study report. Tables, Listings and Figures are numbered following the ICH structure. Table headers, variables names and footnotes will be modified as needed following data analyses. All descriptive and inferential statistical analyses will be performed using SAS® statistical software Version 9.4 or higher, unless otherwise noted.

## TABLE, LISTING AND FIGURE SHELLS

## **Programming note:**

Put Program Name in the footnote where it is stored, Location of Output stored, and Date and time when the output is generated.

T14.1.1 Summary of Patient's Disposition

| Patients Randomized | Test<br>N = xxx<br>n (%) | Reference<br>N = xxx<br>n (%) | Total<br>N = xxx<br>n (%) |
|---|---|---|---|
| Completed Study | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Terminated Early | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Adverse Event | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Lack of efficacy | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Protocol Deviation | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Pregnancy | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| etc. | ` / | | , |
| Other | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

N= number of patients randomized in that particular group; n= number of patient with data available for that particular group; total % is based on N

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

OUTPUT: L:\DEV\755\71675502\SAS\OUT\XXXX Created on: ddmmmyy hh:mm Page 1 of N

**T14.1.2 Summary of Protocol Deviations** 

| | Test<br>N = xxx<br>n (%) | Reference<br>N = xxx<br>n (%) | Total<br>N = xxx<br>n (%) |
|---|---|---|---|
| Total Patients with Protocol Deviations | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Total Deviations | xxx | XXX | XXX |
| Lost to Follow-up | xxx | XXX | XXX |
| Missed Visit | XXX | XXX | XXX |
| Non-compliance with dosing requirements | XXX | XXX | XXX |
| Outside Visit Window | XXX | XXX | XXX |
| Restricted Medication Use | XXX | XXX | XXX |
| Randomized in Error | XXX | XXX | XXX |
| Other | XXX | XXX | XXX |

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

N= number of patients randomized in that particular group; n= number of patient with data available for that particular group; total % is based on N

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

T14.1.3.1 Summary of Patients Excluded from Efficacy Analysis (Population Determination)

| | Test<br>N = xxx<br>n (%) | Reference<br>N = xxx<br>n (%) | Total<br>N = xxx<br>n (%) |
|---|---|---|---|
| Safety Population | xxx (xx.x) | xxx(xx.x) | xxx (xx.x) |
| Excluded from Safety population | xxx (xx.x) | xxx(xx.x) | xxx (xx.x) |
| PP Population | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Excluded from PP population | xxx (xx.x) | xxx(xx.x) | xxx (xx.x) |
| Inclusion/Exclusion criteria not met | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Non-compliant with dosing requirement | xxx (xx.x) | xxx(xx.x) | xxx (xx.x) |
| Major protocol deviations | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| etc. | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Reference: Elimite™ Cream (permethrin) 5% (Prestium Pharma, Inc.)

N= number of patients randomized in that particular group; n= number of patient with data available for that particular group; total % is based on N

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

T14.1.3.2 Summary of Patients Included in Analysis Population by Study Center

| | | | PP | | | Safety | | |
|---|---|---|---|---|---|---|---|---|
| Site<br>No. | Name | Total<br>Randomized | Test | Reference | Total | Test | Reference | Total |
| XX | XXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |
| XX | XXXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

 $PROGRAM: L: \DEV \755 \71675502 \SAS \PGM \XXXX$ 

Created on: ddmmmyy hh:mm

## T14.1.3.3 Study Timelines (Screened subjects)

| | Trial Timelines |
|--------------------------------|-----------------|
| | Date |
| rst Patient First Visit (FPFV) | mm-DDD-YYYY |
| ast Patient Last Visit (LPLV) | mm-DDD-YYYY |
| rial Duration (Days) | XXX |

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71675502\SAS\OUT\XXXX


T14.1.4 Summary of Demographic Data and Baseline Characteristics (Safety Population)

| | | Test<br>n = xxx<br>n (%) | Reference<br>n = xxx<br>n (%) | Total<br>N = xxx<br>n (%) | P-value |
|---|---|---|---|---|---|
| Age (years) | n | XXX | XXX | XXX | X.XXXX |
| | $Mean \pm SD$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ | |
| | Median | XX.X | XX.X | XX.X | |
| | Range | XX.X - XX.X | XX.X - XX.X | xx.x - xx.x | |
| Age Groups | < 18 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | X.XXXX |
| | 18 - 40 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| | 41 - 64 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| | 65 - 75 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| | > 75 | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| Race | American Indian or Alaska Native | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | X.XXXX |
| | Asian | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| | Black/African American | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| | Native Hawaiian or other Pacific<br>Islander | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| | White | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| | Other | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| Ethnicity | Hispanic or Latino | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | X.XXXX |
| | Not Hispanic or Latino | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |

Reference: Elimite™ Cream (permethrin) 5% (Prestium Pharma, Inc.)

N= number of patients randomized in that particular group; n= number of patient with data available for that particular group; total % is based on N

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

**T14.1.4 Summary of Demographic Data** (Safety Population)

| | | Test<br>N = xxx<br>n (%) | Reference<br>N = xxx<br>n (%) | Total<br>N = xxx<br>n (%) | P-value |
|---|---|---|---|---|---|
| Sex | Female | xxx(xx.x) | xxx (xx.x) | xxx (xx.x) | X.XXXX |
| | Male | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| Baseline Severity Score of Nocturnal Itching Pretreatment | None | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | X.XXXX |
| | Mild | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| | Moderate | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| | Severe | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| Baseline Severity of Lesion Count Infestation Pretreatment | Mild | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | x.xxxx |
| | Moderate | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |
| | Severe | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | |

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

N= number of patients randomized in that particular group; n= number of patient with data available for that particular group; total % is based on N

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

OUTPUT: L:\DEV\755\71675502\SAS\OUT\XXXX Created on: ddmmmyy hh:mm Page 1 of N

Similar tables will be created for T14.1.5.

T14.1.5 Summary of Demographic Data (Per-Protocol Population)

T14.1.6 Summary of Microscopic Evaluation of Scabies (Per-Protocol Population)

| Visit | Microscopic<br>Evaluation | Statistic | Test<br>N = xxx<br>n (%) | Reference<br>N = xxx<br>n (%) |
|---|---|---|---|---|
| 1 (Baseline) | Microscopic examination result | Positive | xxx (xx.x) | xxx (xx.x) |
| , | • | Negative | xxx (xx.x) | xxx (xx.x) |
| | Number of scraped sites | n | XXX | XXX |
| | • | Mean $\pm$ SD | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ |
| | | Median | XX.X | XX.X |
| | | Range | XX.X - XX.X | xx.x - xx.x |
| 2 | Microscopic examination result | Positive | xxx (xx.x) | xxx (xx.x) |
| | • | Negative | xxx (xx.x) | xxx (xx.x) |
| | Number of scraped sites | n | XXX | XXX |
| | _ | Mean $\pm$ SD | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ |
| | | Median | XX.X | XX.X |
| | | Range | XX.X - XX.X | xx.x - xx.x |
| 3 (EOS) | Microscopic examination result | Positive | xxx (xx.x) | xxx (xx.x) |
| , , | • | Negative | xxx (xx.x) | xxx (xx.x) |
| | Number of scraped sites | n | XX | XX |
| | - | Mean $\pm$ SD | $xx.x \pm xx.x$ | $xx.x \pm xx.x$ |
| | | Median | XX.X | XX.X |
| | | Range | XX.X - XX.X | XX.X - XX.X |

Reference: Elimite™ Cream (permethrin) 5% (Prestium Pharma, Inc.)

N= number of patients randomized in that particular group; n= number of patient with data available for that particular group; total % is based on N

 $PROGRAM: L: \DEV\755\71675502\SAS\PGM\XXXX$ 

Created on: ddmmmyy hh:mm

T14.1.7 Summary of Frequency of Scabies Signs and Symptoms Rating (Per-Protocol Population)

| | | Test | Reference |
|-------|-----------------------|------------|------------|
| Visit | Grade (Lesion Count) | N = xxx | N = xxx |
| | | n (%) | n (%) |
| 1 | Mild (<50) | xxx (xx.x) | xxx (xx.x) |
| | Moderate $(50 - 100)$ | xxx (xx.x) | xxx (xx.x) |
| | Severe (>100) | xxx (xx.x) | xxx (xx.x) |
| 2 | Mild (<50) | xxx (xx.x) | xxx (xx.x) |
| | Moderate $(50 - 100)$ | xxx (xx.x) | xxx (xx.x) |
| | Severe (>100) | xxx (xx.x) | xxx (xx.x) |
| 3 | Mild (<50) | xxx (xx.x) | xxx (xx.x) |
| | Moderate $(50 - 100)$ | xxx (xx.x) | xxx (xx.x) |
| | Severe (>100) | xxx (xx.x) | xxx (xx.x) |

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

N= number of patients randomized in that particular group; n= number of patient with data available for that particular group; total % is based on N

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX Created on: ddmmmyy hh:mm

T14.1.8.1 Summary of Equivalence Analysis Results of Primary Efficacy Endpoint
(Proportion of Patients in each Treatment Group with Therapeutic Cure (Parasitological Cure plus Clinical Cure)
of Scabies at Day 28 ± 4)
(Per-Protocol Population)

| | | | | Difference Betw | veen Treatments |
|---|---|---|---|---|---|
| Treatment<br>Group | Number of Patients (N) | Number of Patients with<br>Therapeutic Cure (n) | Proportion of Therapeutic Cure (%) | Difference (%) | 90% CI Evaluation |
| Test | Xxx | XXX | XX.X | | |
| Reference | Xxx | XXX | XX.X | XX.X | xx.x - xx.x |

Reference: Elimite<sup>™</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71675502\SAS\OUT\XXXX Page 1 of N

T14.1.8.2 Sensitivity Analysis Summary of Equivalence Analysis Results of Primary Efficacy Endpoint (Proportion of Patients in each Treatment Group with Therapeutic Cure (Parasitological Cure plus Clinical Cure) of Scabies at Day 28 ± 4) (Safety Population)

T14.1.9.1 Supportive Analysis #1: Summary of Equivalence Analysis Results of Primary Efficacy Endpoint (Per-Protocol Population)

| | | • | | Difference Betw | veen Treatments |
|---|---|---|---|---|---|
| Treatment<br>Group | Number of Patients (N) | Number of Patients with<br>Therapeutic Cure (n) | Proportion of Therapeutic Cure (%) | Difference (%) | 90% CI Evaluation |
| Test | Xxx | XXX | XX.X | | |
| Reference | Xxx | XXX | XX.X | XX.X | xx.x - xx.x |

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

The primary analysis will be performed including patients who completed Visit 2 within  $14 \pm 2$  days and Visit 3 within  $28 \pm 4$  days.

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71675502\SAS\OUT\XXXX Page 1 of N

## T14.1.9.2 Supportive Analysis #2: Summary of Equivalence Analysis Results of Primary Efficacy Endpoint (Per-Protocol Population)

Note: The primary analysis will be performed including patients who completed Visit 2 within  $14 \pm 2$  days and Visit 3 between Day 26 and Day 32, inclusive.

# T14.1.9.3 Supportive Analysis #3: Summary of Equivalence Analysis Results of Primary Efficacy Endpoint (Per-Protocol Population)

Note: The primary analysis will be performed including patients who completed Visit 2 within  $14 \pm 2$  days and Visit 3 within  $28 \pm 2$  days.

T14.1.10 Summary of Frequency of Patient Pruritus Assessment (Per-Protocol Population)

| - | | Test | Reference |
|---|---|---|---|
| Visit | Grade (Score) | N = xxx | N = xxx |
| | | n (%) | n (%) |
| 1 | NONE: Complete absence of itching (0) | xxx (xx.x) | xxx (xx.x) |
| | MILD: Slight itching, no sleep loss (1) | xxx(xx.x) | xxx (xx.x) |
| | MODERATE: Definitely present, interrupts sleep (2) | xxx (xx.x) | xxx (xx.x) |
| | SEVERE: Marked, intense, cannot sleep (3) | xxx (xx.x) | xxx (xx.x) |
| 2 | NONE: Complete absence of itching (0) | xxx (xx.x) | xxx (xx.x) |
| | MILD: Slight itching, no sleep loss (1) | xxx (xx.x) | xxx (xx.x) |
| | MODERATE: Definitely present, interrupts sleep (2) | xxx (xx.x) | xxx (xx.x) |
| | SEVERE: Marked, intense, cannot sleep (3) | xxx (xx.x) | xxx (xx.x) |
| 3 | NONE: Complete absence of itching (0) | xxx (xx.x) | xxx (xx.x) |
| | MILD: Slight itching, no sleep loss (1) | xxx (xx.x) | xxx (xx.x) |
| | MODERATE: Definitely present, interrupts sleep (2) | xxx (xx.x) | xxx (xx.x) |
| | SEVERE: Marked, intense, cannot sleep (3) | xxx (xx.x) | xxx (xx.x) |

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

N= number of patients randomized in that particular group; n= number of patient with data available for that particular group; total % is based on N

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX Created on: ddmmmyy hh:mm

# T14.1.11 Overall Summary of Adverse Events (Safety Population)

| Description | Test | Reference | Total |
|---|---|---|---|
| Subjects in Safety Analysis Set | XXX | XXX | XXX |
| Subjects with at least one AE | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Discontinued study drug due to above AE | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| AEs reported | xxx | xxx | XXX |
| Mild | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Moderate | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Severe | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Not Related | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Related | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Death | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Serious AE | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite™ Cream (permethrin) 5% (Prestium Pharma, Inc.)

Note: subjects having multiple AEs within same system organ class were counted only once in respective system organ class. Under any event subjects having multiple AEs with same Preferred Term were counted only once within the respective preferred term.

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX Created on: ddmmmyy hh:mm

# T14.1.12 Summary of Frequency of Adverse Events by Body System (Safety Population)

| | | | Test<br>= xxx | | erence<br>= xxx | |
|---|---|---|---|---|---|---|
| <b>Body System</b> | Preferred Term | Events | Patients<br>n (%) | Events | Patients<br>n (%) | Fisher's<br>p-value |
| Patients with at least one AE | Total | XX | xxx (xx.x) | XX | xxx (xx.x) | X.XXXX |
| Ear and labyrinth disorders | Ear pain etc. | XX | xxx (xx.x) | XX | xxx (xx.x) | X.XXXX |

etc.

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

N= number of patients in safety population in that particular group; n= number of patient with data available for that particular group; total % is based on N

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX Created on: ddmmmyy hh:mm

## T14.1.13 Summary of Frequency of Adverse Events by Relationship (Safety Population)

| | | Test<br># of Events<br>(N = xxx) | | # o | ference<br>f Events<br>= xxx) |
|---|---|---|---|---|---|
| <b>Body System</b> | Preferred Term | Related<br>n (%) | Not Related<br>n (%) | Related n (%) | Not Related<br>n (%) |
| Total AEs<br>Ear and labyrinth disorders | Total<br>Ear pain<br>Hypoacusis | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) | xxx (xx.x)<br>xxx (xx.x)<br>xxx (xx.x) |

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

N = Total number of events in that particular group group; Percentage is based on total number of events.

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

OUTPUT: L:\DEV\755\71675502\SAS\OUT\XXXX Page 1 of N Created on: ddmmmyy hh:mm

# T14.1.14 Summary of Frequency of Adverse Events by Severity (Safety Population)

| | | Test | | Reference | | | |
|---|---|---|---|---|---|---|---|
| | | | # of Events | | | # of Events | |
| | | | (N = xxx) | | | (N = xxx) | |
| <b>Body System</b> | Preferred Term | Mild<br>n (%) | Moderate<br>n (%) | Severe<br>n (%) | Mild<br>n (%) | Moderate<br>n (%) | Severe<br>n (%) |
| Total AEs | Total | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) |
| Ear and labyrinth disorders | Ear pain | xxx(xx.x) | xxx(xx.x) | xxx(xx.x) | xxx (xx.x) | xxx(xx.x) | xxx (xx.x) |
| | Hypoacusis | xxx(xx.x) | xxx (xx.x) | xxx(xx.x) | xxx (xx.x) | xxx(xx.x) | xxx (xx.x) |

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

N = Total number of events in that particular group group; Percentage is based on total number of events.

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX Created on: ddmmmyy hh:mm

675502\SAS\PGM\XXXX OUTPUT: L:\DEV\755\71675502\SAS\OUT\XXXX Page 1 of N

# T14.1.15 Summary of Frequency of Serious Adverse Events (Safety Population)

| Body System | Preferred Term | Test<br># Events | Reference<br># Events |
|---|---|---|---|
| Injury, poisoning and procedural complications | Alcohol poisoning | XXX | XXX |

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71675502\SAS\OUT\XXXX

# T14.1.16 Summary of Vital Signs (Safety Population)

| Vital Signs | Visit | Statistic | Test<br>N = xxx | Reference<br>N = xxx |
|---|---|---|---|---|
| Systolic Blood Pressure (mmHg) | 1 | n | XXX | XXX |
| - | | Mean $\pm$ SD | $xxx.x \pm xx.x$ | $xxx.x \pm xx.x$ |
| | | Median | XXX.X | XXX.X |
| | | Range | xxx.x - xxx.x | xxx.x - xxx.x |
| | 3 | | | |

Diastolic Blood Pressure (mmHg) Pulse Rate (beats/min) Respiration Rate (breaths/min)

Temperature (F)

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite™ Cream (permethrin) 5% (Prestium Pharma, Inc.)

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71675502\SAS\OUT\XXXX

# T14.1.17 Summary of Frequency of Patients with Re-Infestation from Day 14 (treatment success) to Day 28 (treatment failure) (Per-Protocol Population)

| Reference |
|---------------------------------------------------------------------|
| $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ $\mathbf{n} \ (\%)$ |
| XXX (XX.X) |

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

N= number of patients randomized in that particular analysis group; n= number of patient with data available for that particular group; total % is based on N

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71675502\SAS\OUT\XXXX


# T14.1.18 Summary of Frequency of Patients who are Therapeutic Failures on Day $14 \pm 4$ (Per-Protocol Population)

| Test | Reference |
|---|---|
| $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ | $(\mathbf{N} = \mathbf{x}\mathbf{x}\mathbf{x})$ |
| n (%) | n (%) |
| xxx (xx.x) | xxx (xx.x) |

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

N= number of patients randomized in that particular analysis group; n= number of patient with data available for that particular group; total % is based on N

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

11/2/2017 ■ Encube Ethicals ■ 


# L16.2.1 Listing of Discontinued Patients

| Treatment<br>Group | Patient<br>Randomization<br>Number | Discontinuation<br>Reason | Population |
|---|---|---|---|
| Test | XXXX | Withdrawal by Patient | Per-Protocol |
| | XXXX | Lost to Follow-up | Safety |

Reference

Test: Permethrin Cream, 5%, (Encube Ethicals)
Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX


# **L16.2.2** Listing of Protocol Deviations

| Treatment<br>Group | Patient<br>Randomization<br>Number | <b>Event Description</b> | Population |
|---|---|---|---|
| Test | XXXX | Outside Visit Window (Visit 3) | Safety |

Reference

11/2/2017

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

■ Encube Ethicals ■ 

# L16.2.3 Patients Excluded from the Per-Protocol Population

| Treatment<br>Group | Patient<br>Randomization<br>Number | Exclusion Reason |
|---|---|---|
| Test | XXXX | Major protocol deviation |

Reference

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71675502\SAS\OUT\XXXX

# L16.2.4.1 Listing of Demographic Data

| Treatment<br>Group | Patient<br>Randomization<br>Number | Age | Sex | Ethnicity | Race |
|---|---|---|---|---|---|
| Test | XXXX | 30 | Female | Not Hispanic or Latino | Black or African American |

Reference

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

OUTPUT: L:\DEV\755\71675502\SAS\OUT\XXXX Created on: ddmmmyy hh:mm Page 1 of N

# L16.2.4.2 Listing of Medical History

| Treatment<br>Group | Patient<br>Randomization<br>Number | System | Diagnosis or<br>Surgical<br>Procedure | Start Date | End Date | Ongoing |
|---|---|---|---|---|---|---|
| Test | XXXX | Gynecologic | Menopause | yyyy-mm-dd | yyyy-mm-dd | |

Reference

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71675502\SAS\OUT\XXXX


# L16.2.4.3 Listing of Concomitant Medication

| Treatment<br>Group | Patient<br>Randomization<br>Number | Treatment<br>Area | Medication | Dosage | Frequency | Route | Start/End<br>Date/ Ongoing | Indication |
|---|---|---|---|---|---|---|---|---|
| Test | XXXX | No | Lisinopril | 20 MG | QD | РО | yyyy-mm-dd /<br>yyyy-mm-dd | Hypertension |

Reference

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX


# L16.2.4.4 Listing of Treatment for Family Members/Close Contacts

| Treatment<br>Group | Patient<br>Randomization<br>Number | Visit<br>Date | How many members in the patient's house-hold (e.g., close personal contacts, and/or family member(s)) are affected with scabies? | Has the patient come into contact with the affected family member(s) and/or close personal contacts? | Have affected family<br>member(s)/close personal<br>contacts of the patient been<br>given prescription generic<br>permethin? |
|---|---|---|---|---|---|
| Test | XXXX | vvvv-mm-dd | XXX | Yes | Yes |

Reference

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

# L16.2.5.1 Listing of Visit Date Information

| Treatment<br>Group | Patient<br>Randomization<br>Number | Informed<br>Consent Signed | Date Assent<br>Signed | Visit 1 | Visit 2 | Visit 3 /<br>Early<br>Termination | Safety<br>Population | Per-Protocol<br>Population |
|---|---|---|---|---|---|---|---|---|
| Test | XXXX | yyyy-mm-dd | yyyy-mm-dd | yyyy-mm-dd | yyyy-mm-dd | yyyy-mm-dd | Yes | No |

Reference

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71675502\SAS\OUT\XXXX


#### L16.2.5.2 Listing of Drug Administration

| Treatment<br>Group | Patient<br>Randomization<br>Number | Date of<br>First Dose | Date of<br>Last Dose | Total<br>Doses Applied | Treatment<br>Compliance* |
|---|---|---|---|---|---|
| Test | XXXX | yyyy-mm-dd | yyyy-mm-dd | XX | Yes |

Reference

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

 $PROGRAM: L: \DEV \755 \71675502 \SAS \PGM \XXXX$ 

<sup>\*</sup>Treatment compliance will be calculated based off the following criteria: 1.) all patients randomized will have at least 1 dose, confirmed from the study drug administration form via the eCRF. Date of first and last dose and total confirmed doses applied will confirm treatment use. 2.) A patient who is required to dose a second time, compliance will be calculated using criteria 1 and the following data points (via the eCRF) positive microscopic result at Visit 2 and selection of "yes" regarding the question "based on your assessment and microscopic results, is continued treatment required?"

# L16.2.6.1 Listing of Scabies Signs and Symptoms Rating and Microscopic Evaluation of Scabies

| Treatment | Patient | | Scabies | Are there any | Have all | Number | Microscopic | | Parasito- | |
|---|---|---|---|---|---|---|---|---|---|---|
| Group | Randomization | Visit | Lesion | new lesions | original lesions | - | | Clinical | logical | Therapeutic |
| | Number | | Count | present? | healed? | sites | Result | Cure | Cure | Cure |
| Toat | ******* | 1 | Madarata | NIA | NA | 3 | Positive | | | |
| Test | XXXX | 1 | Moderate | NA | | | (mites, eggs) | | | |
| | | 2 | Mala | Ma | No | 3 | Positive | | | |
| | | 2 | Mild | No | | | (eggs) | | | |
| | | 3 | Mild | No | Yes | 0 | Negative | Yes | Yes | Yes |
| | | xx 1 | Moderate NA | NIA | NA | 3 | Positive | | | |
| | XXXX | | | IA | | (eggs) | | | | |
| | | • | 2 Mild | No | No | 3 | Positive | | | |
| | | 2 | | | | | (eggs) | | | |
| | | 3 | Mild | Yes | Yes | 0 | Negative | No | Yes | No |

#### Reference

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

 $PROGRAM: L: \DEV \755 \71675502 \SAS \PGM \XXXX$ 

Created on: ddmmmyy hh:mm

 $OUTPUT: L: \DEV\755\71675502\SAS\OUT\XXXX$ 


# L16.2.6.2 Listing of Patient Pruritus Assessment

| Treatment<br>Group | Patient<br>Randomization<br>Number | Visit 1 | Visit 2 | Visit 3 / Early<br>Termination | No Itch<br>Persistence |
|---|---|---|---|---|---|
| Test | XXXX | 1 (Mild) | 1 (Mild) | 0 (None) | Yes |
| | | 2 (Moderate) | 1 (Mild) | 1 (Mild) | No |

Reference

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite™ Cream (permethrin) 5% (Prestium Pharma, Inc.)

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX


# L16.2.6.3 Listing of Investigator Evaluator Initials On Scabies Signs & Symptoms Rating

| Treatment<br>Group | Randomization | | Visit 2 | Visit 3 / Early<br>Termination |
|---|---|---|---|---|
| Test | XXXX | XYZ | D-G | D-G |

Reference

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

# L16.2.7 Listing of Adverse Events by Treatment

| Treatment<br>Group | Patient<br>Randomization<br>Number | Body System /<br>MedDRA Term /<br>AE Term | Treatment<br>Area | Start /End<br>Date/<br>Ongoing | Severity | Relationship<br>to Study<br>Drug | Outcome | Action Taken/<br>Other Action<br>Taken | SAE | TEAE |
|---|---|---|---|---|---|---|---|---|---|---|
| Test | xxxx | Nervous system disorders / | No | yyyy-mm-dd / | Mild | Related | Recovere | Dose Not | No | Yes |
| | | Headache / | | yyyy-mm-dd | | | d | Changed/ | | |
| | | Headache | | | | | | None | | |

Reference

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71675502\SAS\OUT\XXXX Page 1 of N

11/2/2017 ■ Encube Ethicals ■ 

# L16.2.8.1 Listing of Pregnancy Test Results

| Treatment<br>Group | Patient<br>Randomization<br>Number | Visit 1 | Visit 3 / Early<br>Termination |
|---|---|---|---|
| Test | XXXX | Negative | Negative |

Reference

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm


OUTPUT: L:\DEV\755\71675502\SAS\OUT\XXXX

# L16.2.8.2 Listing of Vital Signs

| Treatment<br>Group | Patient<br>Randomization<br>Number | Visit | Systolic BP (mmHg) | Diastolic BP<br>(mmHg) | Pulse Rate<br>(beats/min) | Respiration<br>Rate<br>(breaths/min) | Temperature (F) |
|---|---|---|---|---|---|---|---|
| Test | XXXX | 1 | 120 | 70 | 84 | 18 | 98.6 |
| | | 3 | 140 | 100 (NCS) | 74 | 18 | 97.0 |

Reference

Test: Permethrin Cream, 5%, (Encube Ethicals)

Reference: Elimite<sup>TM</sup> Cream (permethrin) 5% (Prestium Pharma, Inc.)

PROGRAM: L:\DEV\755\71675502\SAS\PGM\XXXX

Created on: ddmmmyy hh:mm

OUTPUT: L:\DEV\755\71675502\SAS\OUT\XXXX Page 1 of N

11/2/2017 ■ Encube Ethicals ■ 

F15.1.1 Histogram of Proportion of Patients with Therapeutic Cure on Day 28 ±4



#### Reference:

1. FDA Draft Guidance on Malathion, June 2012.